CLINICAL TRIAL: NCT03873792
Title: Oral Probiotics to Allergic Pregnant Mother and Their Offspring to Prevent Allergic Disease
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulties in recruiting participants.
Sponsor: China Medical University Hospital (Other)
Responsible Party: Principal Investigator, Hung-Chih Lin, Attending physician, China Medical University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: CMUH106-REC1-152
Record Dates: First submitted 2019-03-04; First posted 2019-03-13 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Allergic Diseases
Keywords: Allergic diseases; Probiotics; Immunoglobulin E; Intestinal microbiota

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Allergy pregnant women (Other)
  Interventions: Diagnostic Test: Physician diagnoses a history of asthma or eczema or allergic rhinitis or health pregnant women
- Health pregnant women (Other)
  Interventions: Diagnostic Test: Physician diagnoses a history of asthma or eczema or allergic rhinitis or health pregnant women

INTERVENTIONS:
Diagnostic Test: Physician diagnoses a history of asthma or eczema or allergic rhinitis or health pregnant women — Physician diagnoses a history of asthma or eczema or allergic rhinitis

SUMMARY:
The aim of the study is first to detect the difference of the intestinal microbiome between allergic pregnant mother and the non-allergic pregnant mother using the next generation sequence, all postnatal infants will collect the first meconium and feces from one, two, six months to one year old for the same test. The second stage of the study is to restore the allergic pregnant mother abnormal intestinal microbiome with probiotics trying to reduce the incidence of allergic disease of their offspring.

DETAILED DESCRIPTION:
Allergic diseases are the largest group of non-communicable diseases (NCD) with an increasing prevalence in both the developed and developing world. There are significant bodies of research trying to examine the use of probiotics to prevent allergic disease. Though clinical randomized controlled trials and meta-analyses shows benefits of using probiotic supplements during pregnancy and early infant life to prevent the development of atopic dermatitis ; however, Cochrane review found that the benefit is not significant for immunoglobulin E (IgE) associated atopy. The lack of effectiveness that probiotics supplement to prevent allergic offspring to the allergic pregnant mother might due to too late to give probiotics and not give the appropriate probiotics. Investigators speculate that intestinal microbiota of allergic pregnant mother is different from the non-allergic pregnant mother. According to the theory that intestinal microbiome of pregnant mother might affect the offprint's intestinal microbiota during labor and further induce the allergic status.

The aim of the study is first to detect the difference of the intestinal microbiome between allergic pregnant mother and the non-allergic pregnant mother using the next generation sequence, all postnatal infants will collect the first meconium and feces from one, two, six months to one year old for the same test. The second stage of the study is to restore the allergic pregnant mother abnormal intestinal microbiome with probiotics trying to reduce the incidence of allergic disease of their offspring.

Allergic pregnant women who intend to breast- feed their infant are eligible to be enrolled in the study if she has a history of asthma or eczema treated or allergic rhinitis treated by a doctor. All infants born in the study are eligible for inclusion in study outcomes. Study probiotics containing Lactobacillus and Bifidobacterium, and the placebo capsules are made from glucose, both are manufactured by Taiwan Company. After inform consent, probiotics will give to the allergic pregnant women till delivery and infants will have probiotics for 6 months after born. Primary outcome is the prevalence of physician diagnosis atopic eczema and frequency of wheezing attack at 24 month of age.

Randomization is managed by computer at pharmacy of CMUH and concealed from all study staff and participants. An intention-to-treat analysis will be used to assess the effect of probiotics on the 24 month cumulative prevalence of eczema and SCORAD ≥10 using hazard ratios from a Cox's proportional hazards model, and the point prevalence of atopy at age 24 months using relative rates and a chi- squared test. Chi-square test will also be used to compare the proportion in each study group with detectable levels of immunological markers in breast milk. If the data is not log-normally distributed a Wilcoxon Rank-Sum test will be used. Reasons for withdrawal from the study will be recorded and examined for differences between study groups. Adjustment will be made for differences in antibiotic use between study groups. SAS version 9.4 will be used.

ELIGIBILITY:
Inclusion Criteria:

* An adult pregnant mother who is over 20 years old and has a history of asthma or eczema or allergic rhinitis who is exercising autonomous consent.
* Pregnant women over 20 years old without allergies.
* Infants ≧ 37 weeks gestational age.

Exclusion Criteria:

* Under 20 years old.
* Pregnant mothers and babies with congenital immune diseases.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from intestinal microbiome diversity between allergic pregnant mother and the non-allergic pregnant mother. | An average of 2 years for analysis of intestinal microbiome proportion such as Lactobacillus, Bifidobacterium and other genuses.
  To detect the difference of the intestinal microbiome between allergic pregnant mother and the non-allergic pregnant mother using the next generation sequence (NGS).
Change from intestinal microbiome diversity between Infants born from allergic pregnant mothers or non-allergic pregnant mother. | An average of 2 years for analysis of intestinal microbiome proportion such as Lactobacillus, Bifidobacterium and other genuses.
  To detect the difference of the intestinal microbiome between Infants born from allergic pregnant mothers or non-allergic pregnant mother using the NGS.
Change from intestinal microbiome diversity between Infants three months after birth from allergic pregnant mothers or non-allergic pregnant mother. | An average of 2 years for analysis of intestinal microbiome proportion such as Lactobacillus, Bifidobacterium and other genuses.
  To detect the difference of the intestinal microbiome between Infants three months after birth from allergic pregnant mothers or non-allergic pregnant mother using the NGS.
Change from intestinal microbiome diversity between Infants six months after birth from allergic pregnant mothers or non-allergic pregnant mother. | An average of 2 years for analysis of intestinal microbiome proportion such as Lactobacillus, Bifidobacterium and other genuses.
  To detect the difference of the intestinal microbiome between Infants six months after birth from allergic pregnant mothers or non-allergic pregnant mother using the NGS.
Change from intestinal microbiome diversity between Infants one year old after birth from allergic pregnant mothers or non-allergic pregnant mother. | An average of 2 years for analysis of intestinal microbiome proportion such as Lactobacillus, Bifidobacterium and other genuses.
  To detect the difference of the intestinal microbiome between Infants one year old after birth from allergic pregnant mothers or non-allergic pregnant mother using the NGS.
Change from intestinal microbiome diversity between Infants two year old after birth from allergic pregnant mothers or non-allergic pregnant mother. | An average of 2 years for analysis of intestinal microbiome proportion such as Lactobacillus, Bifidobacterium and other genuses.
  To detect the difference of the intestinal microbiome between Infants two year old after birth from allergic pregnant mothers or non-allergic pregnant mother using the NGS.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Pediatrics, Children Hospital, China Medical University, Taichung, Taiwan